CLINICAL TRIAL: NCT00580294
Title: A Pilot Study of Rapid Opioid Rotation and Titration of Oxymorphone
Brief Title: A Pilot Study of Switching From One Pain Medication to Another (Opioid Rotation)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 07-0464
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Pain
Keywords: Sciatica; Diabetic Neuropathies; Complex Regional Pain Syndromes; Low Back Pain; Neck Pain; Headache; Back Pain; Arthritis; Brachial Plexus Injury (stinger/burner); Chronic Pain; Contractures; Diabetes; Fibromyalgia; Foot Pain; Fracture; Hip; Herpes Zoster (shingles); Migraine; Neuropathic Pain; Osteoarthritis; Osteoporosis; Rheumatoid Arthritis; Scoliosis; Nerve pain; Opana; Opioid; Opioid Rotation; Oxymorphone; Morphine; neuropathic; oxycodone
MeSH Terms: conditions — Pain; Sciatica; Diabetic Neuropathies; Complex Regional Pain Syndromes; Low Back Pain; Neck Pain; Headache; Back Pain; Arthritis; Chronic Pain; Contracture; Diabetes Mellitus; Fibromyalgia; Fractures, Bone; Herpes Zoster; Migraine Disorders; Neuralgia; Osteoarthritis; Osteoporosis; Arthritis, Rheumatoid; Scoliosis | interventions — Oxymorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oxymorphone (Experimental): participants switched to oxymorphone extended release (ER) via both oral and intravenous patient-controlled analgesia (IV-PCA) oxymorphone. After 24 hours, participants were discharged with oral oxymorphone ER and oxymorphone immediate release (IR) as needed
  Interventions: Drug: Oxymorphone

INTERVENTIONS:
Drug: Oxymorphone — IV PO
  Other Names: Oxymorphone PO; Oxymorphone IV

SUMMARY:
The purpose of this study is to see if changing from one pain medication like morphine or oxycodone to another pain medication, oxymorphone (OPANA®), will be helpful to patients. This study will examine if the switching from one pain medication to another can be done over a 24 hour period. Oxymorphone, the drug being studied, is an FDA approved drug for treatment of severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to no upper limit
* Chronic pain of nociceptive, neuropathic, or mixed origin
* Patients with chronic non cancer pain
* Ongoing chronic opioid treatment with either oral morphine or oxycodone (long term - more than 3 months of at least a total daily opioid dose of 60 mg morphine or of 30 mg oxycodone)
* Pain of moderate intensity (>4, on the numerical scale 0-10) despite ongoing opioid therapy>
* Non-pregnant, non-lactating women
* Sufficient language skills to communicate with research staff

Exclusion Criteria:Non-ambulatory patients

* Clinically significant respiratory, renal, hepatic, or cardiac disease.
* Documented diagnosis of sleep apnea (the study physician may exclude patients who present with clinical features and complaints suggestive of a diagnosis of probable sleep apnea)
* History of illicit drug or alcohol dependence or abuse, abnormal drug taking / seeking behaviors
* Severe depression (> 26 on the BDI)
* Patients who exhibit a score on the Mini Mental Status Exam (MMSE) of 26 or less. (The range of scores for mild dementia is 21-26 on the MMSE).
* Workman compensation, current or pending medical-legal litigation
* Hypersensitivity to study medication (oxymorphone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pappagallo, MD, Principal Investigator — Icahn School of Medcine at Mount Sinai
Locations (1):
- Icahn School of Medcine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Korkmazsky M, Ghandehari J, Sanchez A, Lin HM, Pappagallo M. Feasibility study of rapid opioid rotation and titration. Pain Physician. 2011 Jan-Feb;14(1):71-82. PMID 21267044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: study conducted at Mount Sinai School of Medicine, Department of Anesthesiology, Clinical Research Center (CRC), New York, NY, and enrolled patients from August 10, 2007 to August 9, 2008
Period: Overall Study
Arm/Group | Oxymorphone
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Oxymorphone: oral oxymorphone ER as the basal opioid during the first 24 hours and supplemental IV-PCA oxymorphone as needed during period 1. During period 2, participants underwent a 2-week oral titration. The oxymorphone ER and IR dosages were adjusted up or down as needed to maintain pain control.
Arm/Group | Oxymorphone
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Average Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Brief Pain Inventory average daily pain (0= no pain, 10=worst imaginable pain)
  units on a scale | 7.34 (1.18)

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Global Impression of Change
Description: PGIC score - participants answered 2 questions regarding change in overall status and overall activity from baseline using a 7-point scale (1 = Very Much Improved, 2 = Much Improved, 3 = Minimally Improved, 4 = No Change, 5 = Minimally Worse, 6 = Much Worse, 7 = Very Much Worse)
Time Frame: baseline and 12 hours
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Oxymorphone
Number analyzed (Participants) | 12
units on a scale | 0.19 [0.08 to 0.44]

2. Primary Outcome: Brief Pain Inventory
Time Frame: Assessed daily for 10 days prior to IV PCA treatment, and assessed daily for 2 weeks after IV PCA treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Oxymorphone
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
This was a pilot open-label study in a small number of participants. A larger randomized study with long-term follow-up and comparison to traditional protocols is necessary to affirm safety. (12 pts had 6 different chronic non-cancer pain diagnoses.)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes